CLINICAL TRIAL: NCT01684228
Title: Impact of Hemodialysis on Exhaled Volatile Organic Compounds in End Stage Renal Disease
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0271-10-RMB-CTIL
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: End Stage Renal Disease
Keywords: End stage renal disease; hemodialysis; breath test; volatile organic compound; dialysis adequacy
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — exhaled breath
Oversight: Data Monitoring Committee: No

SUMMARY:
End stage renal disease (ESRD) is a severe clinical state of irreversible loss of endogenous kidney function, shortening life expectancy, if left untreated. In the state of ESRD, over 5000 uremic toxins are accumulated in the body causing dysfunction of various organ systems. The survival of these patients depends on renal replacement therapies, such as hemodialysis (HD), which artificially purifies the blood from toxins. The investigators assume that some of the uremic toxins are also present in the patient's exhaled breath, and could be detected by a non-invasive and highly sensitive test: a NA-NOSE artificial olfactory system. It is based on analysis of volatile organic compounds (VOCs), a novel, non-invasive field in medical diagnostics. The NA-NOSE is made from an array of nanosensors, and was developed by our collaborator Dr. Hossam Haick (Chemical Engineering, Technion).

In the current study, the investigators utilize this technology to identify VOCs in the exhaled breath of dialysis patients, and to characterize certain patterns of expression that could potentially help in future monitoring of HD adequacy. The investigators plan to collect 150 breath samples from patients before and during dialysis, and from healthy subjects. All participants provide a signed informed consent. Subsequently, analysis of samples will be done at Dr. Haick's laboratory, using Gas-Chromatography/Mass-Spectrometry and parameters extracted from each sensor response.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* End stage renal disease receiving hemodialysis

Exclusion Criteria:

* Age under 18
* Pregnancy
* Malignancy
* Infectious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suheir Assady, MD, Ph.D, Principal Investigator — Department of Nephrology, Rambam-Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel